CLINICAL TRIAL: NCT05661045
Title: The Effect of Blood Carboxyhemoglobin Levels on Total Antioxidant (Tas), Total Oxidant(Tos), Hypoxia Inducible Factor-1a (hif1a) During Low-flow and Normal-flow Anesthesia
Status: Completed | Type: Observational
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Vkoksal, Anestesiology, Ataturk Training and Research Hospital
Other Study IDs: B.30.2.ATA.0.01.00/1
Record Dates: First submitted 2022-12-03; First posted 2022-12-22 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Carbon Monoxide Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group DA: In the Group (DA), the standard consisting of electrocardiogram(ECG), peripheral oxygen saturation (Spo2), and non-invasive blood pressure will be monitored.Prior to induction, the first blood sample (To) will be taken for analysis. After induction of anesthesia with propofol and rocuronium, he will be intubated.Anesthesia will be maintained with desflurane (MAC:1), oxygen (50%), air (50%). After a high flow phase of 4 l/min for 10 min, the fresh gas flow will be reduced to 0.6 L/min and fentanyl,rocuronium will be administered intermittently. Patients will be ventilated with a ventilator at a constant tidal volume (kg x 6 mL) and respiratory rate (12/min). At the 1st hour of low flow anesthesia maintenance, a second blood sample (T1) will be taken for analysis. Patients will be awakened at the end of the case. After the recovery room, it will be transferred to the relevant service. A third blood sample (T2) will be taken at the postoperative 24th hour in the service for analysis.
  Interventions: Procedure: low-flow anesthesia
- Group NA: In the Group (NA),the standard consisting of electrocardiogram(ECG), peripheral oxygen saturation (Spo2),non-invasive blood pressure will be monitored.Prior to induction, the first blood sample (To) will be taken for analysis.After induction of anesthesia with propofol and rocuronium, patients will be intubated. Anesthesia will be maintained with desflurane (MAC:1), oxygen (50%), air (50%). After a high flow phase of 4 l/min for 10 min, the fresh gas flow will be reduced to 2.0 L/min and fentanyl, rocuronium will be administered intermittently. Patients will be ventilated with a ventilator at a constant tidal volume (kg x 6 mL) and respiratory rate (12/min). A second blood sample (T1) will be taken for analysis at the 1st hour of normal flow anesthesia maintenance. Patients will be awakened at the end of the case. After the recovery room, it will be transferred to the relevant service. A third blood sample (T2) will be taken at the postoperative 24th hour in the service for analysis

INTERVENTIONS:
Procedure: low-flow anesthesia — Changes in blood carboxyhemoglobin levels as a result of exposure to rebreathing during low-flow anaesthesia.
  Groups: Group DA

SUMMARY:
In contrast to toxic CO concentrations, low-dose CO acts as a signaling molecule and can exert many complex cytoprotective effects. Therefore, the effects of low-dose CO are being investigated and developed as a new treatment method for use in various disease processes. However, these studies are mostly in vivo and in vitro studies and clinical studies have not reached a sufficient number. In this study, the effect of subclinical COHB levels on biomarkers such as TAS, TOS, HIF-1α will be evaluated.

DETAILED DESCRIPTION:
130 patients aged between 18 and 70 with ASA I-II will be included in the study. Patients will be assigned to one of the two study groups in equal numbers using a computerized random numbers table.

In the 1st group (Group DA), the patients will be taken to the operating table. The standard consisting of electrocardiogram (ECG), peripheral oxygen saturation (Spo2), and non-invasive blood pressure will be monitored. Prior to induction, the first blood sample (To) will be drawn for COHB and biochemistry analysis. After induction of anesthesia with propofol and rocuronium, he will be intubated orotracheal. Anesthesia will be maintained with desflurane (MAC:1), oxygen (50%), air (50%). After a high flow phase of 4 l/min for 10 min, the fresh gas flow will be reduced to 0.6 L/min (low flow anaesthesia) and fentanyl and rocuronium will be administered intermittently. Patients will be ventilated with a ring system ventilator with a newly changed absorber at a constant tidal volume (body weight kg x 6 mL) and respiratory rate (12/min). At the 1st hour of low flow anesthesia maintenance, a second blood sample (T1) will be taken for COHB and biochemistry analysis. Patients will be awakened at the end of the case. After the recovery room, it will be transferred to the relevant service. A third blood sample (T2) will be taken from the patients at the postoperative 24th hour in the service for COHB and biochemistry analysis. Blood carboxyhemoglobin (COHB), total antioxidant status (TAS), total oxidant status (TOS), Hypoxia-inducible factor 1α (HIF-1α) values will be calculated.

Patients in group 2 (Group NA) will be taken to the operating table. The standard consisting of electrocardiogram (ECG), peripheral oxygen saturation (Spo2), and non-invasive blood pressure will be monitored. Prior to induction, the first blood sample (To) will be drawn for COHB and biochemistry analysis. After induction of anesthesia with propofol and rocuronium, he will be intubated orotracheal. Anesthesia will be maintained with desflurane (MAC:1), oxygen (50%), air (50%). After a high flow phase of 4 l/min for 10 min, the fresh gas flow will be reduced to 2.0 L/min (normal flow anaesthesia) and fentanyl and rocuronium will be administered intermittently. Patients will be ventilated with a ring system ventilator with a newly changed absorber at a constant tidal volume (body weight kg x 6 mL) and respiratory rate (12/min). A second blood sample (T1) will be taken for COHB and biochemistry analysis at the 1st hour of normal flow anesthesia maintenance. Patients will be awakened at the end of the case. After the recovery room, it will be transferred to the relevant service. A third blood sample (T2) will be taken from the patients at the postoperative 24th hour in the service for COHB and biochemistry analysis. Blood carboxyhemoglobin (COHB), total antioxidant status (TAS), total oxidant status (TOS), Hypoxia-inducible factor 1α (HIF-1α) values will be calculated.

SPSS 25.0 (IBM Corporation, Armonk, New York, United States) program will be used in the statistical analysis of the variables obtained as a result of the study. The conformity of the data to the normal distribution will be evaluated with the Shapiro-Wilk test and the homogeneity of variance with the Levene test. Independent sample t test and Mann Whitney u test will be used to compare two groups with each other according to quantitative data. In order to examine the correlations of the variables with each other, appropriate ones from Pearson Correlation, Kendall's tau-b and Spearman's rho tests will be used considering the distribution of the data. According to the results of the correlation analysis, it will be supported by regression analysis when necessary. Pearson Chi-Square and Fisher Exact tests will be used to compare categorical variables with each other. Quantitative variables will be shown in the tables as mean (standard deviation) and median (Maximum-Minimum), and categorical variables as n(%). Variables will be analyzed at 95% confidence level and p value less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* ASA I-II
* none-smoking
* without systemic disease
* elective surgery with general anesthesia

Exclusion Criteria:

* over 70 years old
* with cardiovascular disease
* with respiratory system disease
* liver or kidney disease
* pregnant or nursing female patient
* those who do not want to participate
* patient with multi-trauma
* ASA III and above
* emergency surgery
* surgery with blood transfusion
* smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-80, without systemic disease, non-smoker, who will undergo elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Cohb | t1: first hour of surgery
  carboxyhemoglobin
tas | t1: first hour of surgery
  total antioxidant status
tos | t1: first hour of surgery
  total oxidant status
hif-1α | t1: first hour of surgery
  hypoxia inducible factor 1α

CONTACTS AND LOCATIONS:
Overall Officials: VEYSEL KOKSAL, PROF ASS, Principal Investigator — same
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bauer I, Pannen BH. Bench-to-bedside review: Carbon monoxide--from mitochondrial poisoning to therapeutic use. Crit Care. 2009;13(4):220. doi: 10.1186/cc7887. Epub 2009 Aug 14. PMID 19691819
- [Result] Lee SJ, Ryter SW, Xu JF, Nakahira K, Kim HP, Choi AM, Kim YS. Carbon monoxide activates autophagy via mitochondrial reactive oxygen species formation. Am J Respir Cell Mol Biol. 2011 Oct;45(4):867-73. doi: 10.1165/rcmb.2010-0352OC. Epub 2011 Mar 25. PMID 21441382